CLINICAL TRIAL: NCT03287895
Title: A Multifaceted Tool to Improve Decision Making About Cardio-Pulmonary Resuscitation (CPR) for Hospitalized Patients Who Are Seriously Ill
Brief Title: Improving Decisions About CPR
Acronym: iCANACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Frailty Network (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20170531
Record Dates: First submitted 2017-08-28; First posted 2017-09-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: CPR Decision-Making
Keywords: Cardio-pulmonary resuscitation; CPR; Decision-making; Advance Care Planning; End of life; Code Status; Goals of Care; Communication
MeSH Terms: conditions — Death; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Decision Support (Experimental): In addition to the regular conversation about CPR that a patient's physician may have with them, participants will be given a two-part intervention. First, the participant will receive a values clarification tool which helps them rate and understand which relevant values are most important to them. There are two forms of this tool, a full and simplified version. All participants in this arm will receive both, in randomized order. The second aspect of the intervention is an educational video about the potential risks and benefits of CPR, which all participants in this arm will receive.
  Interventions: Behavioral: Decision Support
- Control (No Intervention): Participants in this arm will receive usual care, the regular conversation about CPR that their physician may have with them.

INTERVENTIONS:
Behavioral: Decision Support — A two-part intervention to help patients make better decisions about CPR
  Arms: Intervention - Decision Support

SUMMARY:
Objective

The primary objective is to evaluate the efficacy of a multi-faceted, clinical decision support intervention aimed at improving the quality of decisions about Cardio Pulmonary Resuscitation (CPR) for seriously ill, elderly patients in hospital.

The hypothesis is that fewer patients in the intervention group will have a documented order for CPR and they will have greater satisfaction with decision making about CPR than patients in the control group.

DETAILED DESCRIPTION:
Methodological Approach

The study will be a randomized controlled trial comparing a multi-faceted decision support intervention to usual care for hospitalized patients. The primary objective of this study is to determine if our multifaceted intervention changes decisions about CPR. The components of the multifaceted intervention have already been evaluated for feasibility and acceptability in the hospital setting. The intervention has two parts: the first is a values clarification exercise, and the second part is a CPR video decision aid that explains the risks and benefits of CPR as well as the reasons a patient may choose to receive CPR or not. From previous research it is known that many hospitalized patients have prescribed orders for CPR despite expressing a preference not to have CPR when asked. Furthermore patients often have expressed values that are not concordant with their expressed wishes regarding resuscitation. Therefore it is hypothesized that fewer patients in the intervention group will have a documented order for CPR and they will have greater satisfaction with decision making about CPR than patients in the control group.

We will conduct sensitivity analyses to investigate whether the intervention is more effective among patients who remain in hospital longer after enrollment. We will measure the intervention effect among patients who remained in hospital for fewer than three days after enrollment, among patients who were in hospital for 3-7 days after enrollment, and among patients who remained in hospital for longer than 7 days post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible to receive CPR
2. Satisfying at least one of the following criteria groups

   1. 55 years of age or older with one or more of the following diagnoses:

      * Chronic obstructive lung disease (2 of the 3 of: baseline PaCO2 of > 45 torr, cor pulmonale; respiratory failure episode within the preceding year; forced expiratory volume in 1 sec <0.5 L)
      * Congestive heart failure (New York Heart Association class IV symptoms and left ventricular ejection fraction < 25%)
      * Cirrhosis (confirmed by imaging studies or documentation of esophageal varices and one of three conditions; hepatic coma, child's class C liver disease, or child's class B liver disease with gastrointestinal bleeding)
      * Cancer (metastatic cancer or stage IV lymphoma)
      * End-stage dementia (inability to perform all ADLs, mutism or minimal verbal output secondary to dementia, bed-bound state prior to acute illness).
   2. 80 years of age or older and admitted to hospital from the community for an acute medical or surgical condition.
   3. If none of the above criteria are met, any patient whose death within the next 6 months would not surprise any member of their care team.
   4. At least 55 years old and predicted risk of death in the next 12 months of >=10% as calculated with the HOMR Now! Score

Exclusion Criteria:

* Patients or SDMs who do not speak English.
* Patients or SDMs who do not provide informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
CPR Orders | 14 days post enrollment
  The proportion of patients with an order for CPR in the medical record

SECONDARY OUTCOMES:
Patient/Substitute Decision Maker (SDM) satisfaction with decision-making | Immediately after intervention, or enrollment for control group
  Decision-making domain of the Canadian Health Care Evaluation Project (CANHELP) questionnaire
Decisional Conflict | Immediately after intervention, or enrollment for control group
  Measured using a modified version of the Decisional Conflict Scale
Health Resource Usage | From enrolment to 1 year after enrollment.
  Case costing system at the Ottawa Hospital data warehouse used to measure total cost of hospital care for patients (direct and indirect)
Number of documented goals of care conversations | Between study enrollment and up to 14 days post enrollment
  Count of documented goals of care conversations, defined as "a conversation that addressed at least one of the following domains: patient values and goals; prognosis or illness understanding; end-of-life care planning; or code status (that is, whether or not a patient has requested resuscitation in the event of a Code Blue) or desire for other life-sustaining treatments or procedures." (Lakin et al. Health Affairs 36, no.7 (2017):1258-1264). We will report the presence or absence of any goals of care conversation, as well as the mean number of conversations in each group.
Quality of documented goals of care conversations | Between study enrollment and up to 14 days post enrollment
  Mean quality score for the first instance of a goals of care conversation following study enrollment. Quality assessed using the scale developed for Lakin et al. 2017. This scale has a maximum score of 17 and a minimum score of 1.
SDM Self-efficacy | Immediately after intervention, or enrollment for control group
  For substitute decision-makers who participate, their confidence to make medical decisions on behalf of their loved will be measured using a 5-question questionnaire. The questionnaire asks SDMs to rate their knowledge and confidence about different aspects of decision-making, on a scale from 0 (not confident at all) to 4 (very confident). SDM self-efficacy will be calculated as the mean score among the 5 questions.
Number of emergency department visits | In the year following index admission
  Count of presentations to emergency department
Number of participants with in-hospital mortality | In the year following index admission
  Participants will contribute to this measure if they die while admitted to hospital
Discharge Disposition | End of index admission
  Patient destination on discharge from index admission (home, home with support, rehabilitation, long-term care, etc).
Number of hospital admissions | In the year following index admission
  Count of admissions to hospital
Number of hospital days | In the year following index admission
  Count of days admitted to hospital
Number of ICU days | In the year following index admission
  Count of days admitted to an intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kobewka, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital General Campus, Ottawa, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No